CLINICAL TRIAL: NCT01881516
Title: Randomized, Double-Blind, Placebo-Controlled, Stage II Trial of Acupuncture For Lung Cancer Patients With Cancer Related Fatigue（CRF）
Brief Title: Acupuncture Research on Lung Cancer Patients With Cancer Related Fatigue（CRF）
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, xie jing, attending, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIM2013-F
Record Dates: First submitted 2013-06-13; First posted 2013-06-19 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Lung Cancer; Cancer Related Fatigue
MeSH Terms: conditions — Lung Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture (Active Comparator): Participants will receive 30-min sessions of true acupuncture per week after randomization for 6 weeks
  Interventions: Device: acupuncture
- sham acupuncture (Sham Comparator): Participants will receive 30-min sessions of sham acupuncture per week after randomization for 6 weeks.
  Interventions: Device: sham acupuncture

INTERVENTIONS:
Device: acupuncture — once per week for 6 weeks，30 mins for each treatment and for seven main acupoints
  Other Names: Streitberger needles
  Arms: Acupuncture
Device: sham acupuncture — the same acupoints and time as in acupuncture arm, but use a Park Sham Device
  Other Names: Park Sham Device
  Arms: sham acupuncture

SUMMARY:
we plan to conduct this trial to find out：

* If acpuncture treatment could relieve CRF among lung cancer patients receiving chemo- or radio-therapy？
* How about the extent it relieves？the safety and applicability ？
* What's the possible influential factor and mechanism ？

ELIGIBILITY:
Inclusion Criteria:

* Patients who are pathologically/cytologically diagnosed as NSCLC and received radiotherapy with or without chemotherapy, and the last radio- or chemo-therapy must be at least 30 days prior to initiation of experimental treatment;
* Participants who meet the diagnosis criteria of CRF（ICD-10 criteria);
* The first time to receive acupuncture treatment;
* The age is between 18 and 65 years old;
* Mean baseline fatigue as measured by the Brief Fatigue Inventory (BFI) must be four or above;
* ECOG performance status 0, 1 or 2.
* Patients must have adequate organ functions reflected by the laboratory criteria below: neutrophil counts ≥ 1.5×109 /L, platelet count ≥ 100 x 109/L, hemoglobin ≥ 85 g/L, Serum creatinine < 2.0 mg/dL, Bilirubin < 1.5 mg/dL, ALT < 3 x normal, albumin >30g/L.
* Have not taken any hypnotic, melatonin, or antidepressants within 30 days;
* Willing to finish the whole observation period;
* With written consent form signed by themselves.

Exclusion Criteria:

* Participants in other clinical research;
* Can not be pathologically or cytologically diagnosed as NSCLC;
* ECOG 3~4;
* Pregnant woman;
* >65 or <18 years old;
* Patients with evidence of any cognitive dysfunction that would limit their abilities to report fatigue;
* Patients who have received acupuncture ever before;
* Received surgery, immunotherapy or target therapy within one month before the recruition；
* Taking warfarin or heparin, a bleeding tendency exists;
* Infection, ulceration or hyperalgesia at or near the local acupoints' skin，or with active infections；
* There are cerebral vascular accident history or spinal cord injury history；
* Combination with other serious diseases or condition, including congestive heart failure, Unstable angina pectoris, myocardial infarction during the past six months, serious's arrhythmia, mental disorders, drug abuse, etc.;
* Patients with a life expectancy < 3 months;
* Patients with a past history of therapy or scheduled visits non-compliance, as determined by their treating physician.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Brief Fatigue Inventory, BFI | 12 months

SECONDARY OUTCOMES:
MDASI-C | 12 months
number of adverse events of acupuncture | 24 months
FACT-L | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: jing xie, MD, Principal Investigator — Fudan University; zhen chen, MD, Study Director — Fudan University; qiang zhi meng, MD, Study Chair — Fudan University